CLINICAL TRIAL: NCT07019688
Title: Evaluation of Anxiety During Impacted Molar Extraction: The Influence of Verbal, Traditional, and AI-Generated Information Methods on Anesthesia Management
Brief Title: Anxiety and Information Methods in Molar Extraction
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Gözde Nur Erkan, Assistant Professor, Department of Oral and Maxillofacial Surgery, Kırıkkale University
Other Study IDs: Approval Number: 2025.01.07
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Artifical Intelligence; Health Communication; Information Dissemination; Decision Support Techniques
Keywords: Dental anxiety; Impacted molar extraction; Patient education; Health communication; Artificial intelligence; Anesthesia-related anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Standard Info: Participants receive the standard written information routinely provided before molar tooth extraction.
  Interventions: Other: Standard Information
- Group 2: Clinician Info: Participants receive written information prepared by clinicians that includes answers to the most frequently asked questions from previous patients.
  Interventions: Other: Clinician Information
- Group 3: AI Info: Participants receive written information generated by ChatGPT based on the identified frequently asked questions.
  Interventions: Other: AI Info

INTERVENTIONS:
Other: Standard Information — Participants will receive only the standard written information routinely provided prior to dental procedures. This version does not include any additional content related to frequently asked questions.
  Groups: Group 1: Standard Info
Other: Clinician Information — Participants will receive written information prepared by clinicians, which includes responses to the most frequently asked questions collected from patients undergoing same procedures.
  Groups: Group 2: Clinician Info
Other: AI Info — Participants will receive written information generated by ChatGPT, based on the identified frequently asked questions and formulated specifically for this study.
  Groups: Group 3: AI Info

SUMMARY:
The aim of this clinical study is to investigate the effects of different information methods on patients' anxiety levels during dental procedures under anesthesia. Additionally, the study seeks to evaluate patients' concerns and willingness regarding dental treatment under anesthesia, as well as their awareness of the associated risks.

The main questions this study aims to answer are:

* How do various information methods influence patients' anxiety levels related to dental procedures under anesthesia?
* What is the relationship between patients' anxiety levels and their awareness of risks associated with dental treatment under anesthesia?

The study hypothesizes that different information methods may vary in their effectiveness at reducing patient stress, and that patients' anxiety levels regarding dental treatment under anesthesia may be associated with their knowledge about potential risks.

DETAILED DESCRIPTION:
In this study, questions from 25 patients scheduled for molar tooth extraction will first be collected, and the 20 most frequently asked questions will be identified. The answers to these questions will then be incorporated into routine information procedures. Researchers will prepare verbal, standard written, and written informative materials addressing these questions. To evaluate the impact of artificial intelligence, the identified questions will be submitted to ChatGPT, and the AI-generated responses will be used to create an informational form.

Following the identification of frequently asked questions, newly enrolled patients will be randomly assigned into three groups. Group 1 will receive standard written information, Group 2 will receive clinician-prepared written information containing answers to the identified questions, and Group 3 will receive a written informational form prepared by ChatGPT based on the identified questions. Each group will comprise 35 patients.

Prior to receiving information, participants will complete a baseline survey. Patients will be assigned unique codes, and data including age, gender, educational status, Modified Dental Anxiety Scale (MDAS) scores, and anxiety levels related to dental procedures and anesthesia will be collected. Patients will then receive group-specific information. A follow-up appointment will be scheduled one week later. At this visit, anxiety levels will be reassessed using the MDAS, and additional information will be collected regarding sources consulted for supplementary information (e.g., social media, websites, patient testimonials) and patients' knowledge of anesthesia-related complications. Patients with an MDAS score below 19 will undergo molar tooth extraction under local anesthesia. Those with an MDAS score of 19 or higher will be referred to the anesthesiology faculty member, who also serves as the principal investigator of this study, for the necessary procedures related to dental treatment under anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Indication for moderately difficult, non-complicated impacted mandibular molar extraction
* Aged 18-40 years
* No systemic disease or regular medication use
* No previous procedures under sedation or general anesthesia
* No history of impacted molar surgery or complicated extractions
* No prior verbal, written, or visual information on molar extractions

Exclusion Criteria:

* Complex or multiple (>2) molar extractions
* Intellectual disability
* Emergency cases
* Refusal to participate or to receive preoperative information

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of adult patients aged 18 to 40 years who are scheduled for the extraction of impacted mandibular molar teeth with a predicted moderate level of difficulty and no anticipated complications. Eligible participants must be systemically healthy, not taking any regular medications, and must have no prior history of sedation, general anesthesia, or surgical removal of impacted molars. Individuals who have previously received verbal, written, or visual information regarding impacted molar extraction will be excluded. Only patients who voluntarily consent to participate and are agreeing to receive preoperative information will be included.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Change in Dental Anxiety Level | Baseline (pre-information) and 1 week post-information
  Change in anxiety levels measured using the Modified Dental Anxiety Scale (MDAS) before and one week after the informational intervention. The primary comparison will assess differences between the three groups receiving different information methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Faculty of Dentistry, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The Individual Participant Data (IPD) will not be publicly available but can be shared upon reasonable request.